CLINICAL TRIAL: NCT06915116
Title: Acupuncture for Adolescent and Young Adult Cancer Patients: (AcuAYA)
Brief Title: Acupuncture for People Experiencing Period Loss Due to Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-020
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Period Problem
Keywords: Acupuncture; Stage I cancer; Stage II cancer; Stage III cancer; Period Loss Due to Chemotherapy
MeSH Terms: conditions — Neoplasms; Menstruation Disturbances | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This is a two arm randomized study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Participants in the acupuncture group will receive 12 acupuncture treatments over 12 weeks during the study.
  Interventions: Procedure: Acupuncture
- Wait-list Control (Active Comparator): Participants in the wait-list control group will be put on a wait-list and have the option to receive the same acupuncture treatment as the acupuncture group after a 16-week waiting period
  Interventions: Other: No Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture will be delivered by licensed experienced acupuncturists at MSK. The intervention includes 12 treatments of acupuncture over 12 weeks (i.e. one treatment a week) with a +/- 14-day window. When patients experience menses recovery during the treatment period, they have the option to discontinue treatment or continue receiving up to 12 acupuncture sessions for symptom management over 12 weeks.
  Arms: Acupuncture group
Other: No Acupuncture — Will have the option to receive the same acupuncture treatment as the acupuncture group after a 16-week waiting period
  Arms: Wait-list Control

SUMMARY:
The purpose of this study is to find out whether it is practical (feasible) to use acupuncture to treat period loss (amenorrhea) caused by chemotherapy treatment in people with cancer. The researchers will look at how many participants enroll and complete the study. The researchers will also study how treatment with acupuncture affects the amount of time for the menstrual cycle to return and symptoms and quality of life related to amenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* English speaking women under the age of 40, with a history of stage I, II, or III cancer at the age of 18-39
* Premenopausal status with regular menstruation at the time of diagnosis by patient report
* Completed chemotherapy within the past year
* Report cessation of menses during or after chemotherapy and have not experienced menses recovery at the time of enrollment.
* Have been without menses for at least 3 months following the completion of chemotherapy
* Willing to adhere to all study-related procedures, including randomization to one of the two possible arms: acupuncture and WLC

Exclusion Criteria:

* Metastatic cancer (stage IV)
* Had been pregnant or lactating within 3 months prior to enrollment
* History of hysterectomy or oophorectomy
* Ongoing or planned radiation or surgery within 4 months from randomization
* Use of acupuncture for menses recovery within 3 months of enrollment
* Had been or will be receiving ovarian suppression medicine, such as leuprolide (Lupron) and goserelin (Zoladex), or hormonal contraception drugs within 3 months of enrollment or during the study period

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Menses recovery
Enrollment: 60 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | 1 year
  This is the proportion of patients who enroll in the study among those who are eligible and offered participation. Reason for not participating will be documented (e.g. time/commitment, not wanting to be randomized, does not want the study intervention).
Acupuncture treatment adherence rate. | up to 16 weeks
  adherence rate is the proportion of patients randomized to the Acupuncture arm who are treatment adherent, defined as completing 10 or more of the 12 acupuncture sessions.

SECONDARY OUTCOMES:
Menses recovery | 1 year
  Upon the return of menstruation, participants will inform to their CRCs. The CRCs will then send them the Bleeding Diary which is a link provided through REDCap to record the date and characteristics of their menses. They will be required to fill out this link daily until the menstrual cycle concludes

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm